CLINICAL TRIAL: NCT02640495
Title: A Multicenter, Prospective, Observational Study to Assess the Efficacy of Artesunate in Malaria Treated With Parenteral Artesunate in Areas With Artemisinin Resistance A Study by the Tracking Resistance to Artemisinin Collaboration (TRAC)
Brief Title: Artemisinin Resistance In Malaria Treated With IV Artesunate
Acronym: ARIMTIA
Status: Withdrawn | Type: Observational
Why Stopped: Due to the relative low incidence of severe malaria in Southeast Asia.
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Oxford University Clinical Research Unit, Vietnam (Other)
Responsible Party: Sponsor
Other Study IDs: BAKMAL1504
Record Dates: First submitted 2015-11-16; First posted 2015-12-29 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Malaria
Keywords: Treatment Efficacy; drug resistance; Artemisinin
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study subjects: Patients admitted with malaria, caused by Plasmodium falciparum, treated with parenteral artesunate.
  Interventions: Drug: Intravenous Artesunate as part of standard medical practice

INTERVENTIONS:
Drug: Intravenous Artesunate as part of standard medical practice — Intravenous Artesunate 2.4 mg/kg

SUMMARY:
The spread of artemisinin resistant falciparum malaria presents new challenges to both the control and treatment of malaria. Loss of ring stage susceptibility to the artemisinins might jeopardize the use of parenteral artesunate as the first line drug for the treatment of severe falciparum malaria.

The purpose of this study is to assess the effect of artemisinin resistance (defined by a Kelch13 mutation with known functional significance) in P. falciparum malaria requiring parenteral artesunate treatment on lactate clearance parameters.

DETAILED DESCRIPTION:
The investigators propose a multi-center observational study to assess the effect of artemisinin resistance (as defined by the presence of relevant Kelch13 mutations) on the efficacy of parenteral artesunate for the treatment of malaria, stratified for disease severity on admission.

The patients will receive the standard intravenous treatment for severe malaria (parenteral artesunate). Primary endpoints will be the plasma lactate concentration at 12 hours as a proportion of the plasma lactate at the start of treatment. Secondary endpoints will be improvement of Glasgow or Blantyre Coma Scores and other indicators of neurological recovery or deterioration, parasite clearance rates, time until resolution of fever, development of new severity or neurological signs under treatment, development of severe anemia, renal and hepatic injury, total duration of hospitalization , outcome of pregnancy in pregnant female patients, mortality rates and the necessity to treat with antibiotics, need for renal replacement therapy, mechanical ventilation, blood transfusion and rescue treatments.

On admission blood will be taken for the determination of genetic markers of antimalarial resistance (including Kelch13 mutations of known functional significance) and in vitro sensitivity tests to artemisinins and other antimalarials. Additional blood samples will be used for measuring plasma organic acid biomarkers of severe falciparum malaria measured by mass spectrometry. Difference in the kinetics of these acids will be an additional endpoint. Difference in the transcriptome of p. falciparum will be assessed by RNA measurements at baseline and 3 timepoints during treatment.

The proposed sites in Vietnam and Cambodia have been chosen based on the prevalence of artemisinin resistant falciparum malaria, incidence of severe malaria and local experience in participating in clinical trials.

Interim analysis:

To ensure timely recognition of the effect of artemisinin resistance on the outcome in malaria treated with parenteral artesunate, an interim analysis will be performed after the inclusion of 60 patients or one malaria transmission season (whatever comes first). An independent Data Safety Board will assess whether the difference in outcome between infections with artemisinin resistant versus sensitive strains warrants early termination and reporting of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged over 6 months old
* Acute severe P. falciparum malaria or another indication to treat with IV artesunate. Defined as one or more of the following, occurring in the absence of an identified alternative cause, and in the presence of P. falciparum asexual parasitaemia:

  * Prostration OR obtundation
  * BCS<3 (preverbal children) or GCS<11 (adults)
  * Convulsion in last 24 hours
  * Suspected acidosis, manifesting as acidotic breathing
  * Respiratory distress manifesting clinically (nasal flaring/indrawing) or oxygen saturation <92% or respiratory rate >30/min
  * History of anuria
  * Jaundice and/or hemoglobinuria
  * Hemoglobin <7 g/dl or hematocrit <20%
  * Significant bleeding including recurrent or prolonged bleeding from nose gums or venipuncture sites; hematemesis or melena
  * Shock defined as systolic blood pressure <70 mm Hg (children) OR <80 mm Hg (adults)
  * P. falciparum parasitaemia >10%
  * Indication for parenteral antimalarial treatment (as assessed by clinician) other than nausea and vomiting. These may include laboratory findings such as:

    * Creatinine >2.5 mg/dL (>220uM/L) or blood urea >56mg/dL (>20 mM/L)
    * Glucose <4.0 mmol/L (<72mg/dL)
    * Bilirubin > 3 mg/dL (>50uM/L)
    * Hemoglobin <7g/dL or Hematocrit <20%
    * P. falciparum parasitaemia >4%
    * Venous plasma lactate >5 mM, Base deficit of >8meq/L or bicarbonate <15mM
  * Written informed consent or consent by locally accepted representative in the case of patients rendered incapable of providing consent due to illness

Exclusion Criteria:

* History of 2 or more doses of parenteral antimalarial treatment in the previous 24 hours
* History of allergy or known contraindication to artemisinins

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted with malaria, caused by Plasmodium falciparum, treated with parenteral artesunate.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Absolute reduction of lactate | 12 hours
  Absolute reduction of lactate at 12 hours after the first artesunate treat-ment compared to baseline.

SECONDARY OUTCOMES:
Time needed until a plasma lactate concentration <2 mmol/L | 42 days
Change in Glasgow Coma Score (GCS) or Blantyre Coma Score (BCS) | 12 hours
  at 12 hours after initial treatment and coma recovery time defined as GCS>10 or BCS>3 and GCS=15 and BCS=5
Base excess clearance after 12 hours | 42 days
  Base excess clearance after 12 hours as proportion of the base excess at presentation
Time until a base excess concentration ≥ minus 2 mmol/L | 42 days
Time to resuming the ability to sit, eat, drink, stand unsupported and walk | 42 days
The parasite clearance half-life | 48 hours
The parasite clearance ratios at H28 and H48 compared to parasite count on admission | 48 hours
The parasite clearance time for parasite count to fall to 50%, 90% and 99% of initial parasite density | 7 days
Differences in transcriptome patterns between artemisinin resistant parasites and artemisinin sensitive parasites at baseline | H0
Differences in transcriptome patterns between artemisinin resistant parasites and artemisinin sensitive parasites at H6 | H6
Differences in transcriptome patterns between artemisinin resistant parasites and artemisinin sensitive parasites at H12 | H12
Differences in transcriptome patterns between artemisinin resistant parasites and artemisinin sensitive parasites at H48 | H48
Time until resolution of fever | 14 days
  (time until tympanic temperature first <37.5 Celsius and below 37.5C for 24 h)
Proportion of patients developing new malaria | 42 days
  Proportion of patients developing new malaria severity signs as defined in the 2014 WHO severe malaria guidelines
Proportion of patients developing new neurological signs assessed by neurological examination during hospitalization | 42 days
Prevalence of neurological sequelae assessed by neurological examination at discharge | 42 days
Prevalence of neurological sequelae assessed by neurological examination at day 7 | 7 days
Prevalence of neurological sequelae assessed by neurologicalexamination at day 14 | 14 days
Prevalence of neurological sequelae assessed by neurological examination at day 28 if day 14 is abnormal | 28 days
Prevalence of neurological sequelae assessed by neurological examination at day 42 if day 28 is abnormal | 42 days
Severity of neurological sequelae assessed by neurological examination at discharge | 42 days
Severity of neurological sequelae assessed by neurological examination at day 7 | 7 days
Severity of neurological sequelae assessed by neurological examination at day 14 | 14 days
Severity of neurological sequelae assessed by neurological examination at day 28 if day 14 is abnormal | 28 days
Severity of neurological sequelae assessed by neurological examination at day 42 if day 28 is abnormal | 42 days
Proportion treated with quinine | 42 days
  as a rescue treatment, antibiotics, blood products, anticonvulsants, renal replacement therapy, mechanical ventilation therapy, vasopressive drugs and oxygen therapy
In hospital mortality | 42 days
Day 7, 14 hemoglobin or hematocrit levels | 42 days
  and in addition at day 28 and 42 if abnormal at day 14 or day 28 respectively
Creatinine levels daily | 42 days
  during the first four days and thereafter on day 7 and 14 and in addition on day 28 and 42 if abnormal on day 14 or day 28 respectively
Bilirubin, Alanine transaminase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase levels daily | 42 days
  during the first four days and thereafter on day 7, 14 and in addition on day 28 and 42 if abnormal on day 14 or 28 respectively
Plasma biomarkers of severe (artemisinin resistant) malaria | 42 days
outcome of pregnancy during hospitalization | 42 days
  If pregnant
Time until discharge | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Arjen M Dondorp, MD, Principal Investigator — Mahidol Oxford Research Unit (MORU)